CLINICAL TRIAL: NCT04895644
Title: Duration Of External Neck Stabilisation Following Odontoid Fracture In Older Or Frail Adults: A Randomised Controlled Trial Of Early Versus Late Collar Removal
Brief Title: The Duration of External Neck Stabilisation (DENS) Trial
Acronym: DENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC21022
Record Dates: First submitted 2021-03-31; First posted 2021-05-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Odontoid Fracture
Keywords: Elderly; Hard Collar; Dens; Odontoid

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Hard Collar (Experimental): Patient randomised to not wearing a Hard Collar for 12 weeks
  Interventions: Other: No Hard Collar
- Standard Care Arm - Hard Collar (No Intervention): Patient randomised to wearing a Hard Collar for 12 weeks - standard care

INTERVENTIONS:
Other: No Hard Collar — The patient in the intervention arm will not wear a Hard Collar for 12 weeks post injury
  Arms: No Hard Collar

SUMMARY:
The Duration of External Neck Stabilisation (DENS) study is a randomised controlled trial comparing early removal of a hard collar with treatment in a hard collar for 12 weeks in older or frail adults with odontoid (dens) fractures. The primary outcome measure is QoL assessed using the EQ-5D-5L at 12 weeks following injury. The aim of the study is to determine whether management without a collar improves outcome, compared to management with a collar. Cost efficiency will be assessed over the observed 6 months using standard NICE reference case methodology.

DETAILED DESCRIPTION:
This is a non-blinded randomised controlled trial with nested qualitative research comparing early removal of a hard collar (intervention) with treatment in a hard collar for 12 weeks (standard care) in older or frail adults with odontoid peg fractures. The primary outcome measure is QoL assessed using the EQ-5D-5L at 12 weeks following randomisation.

Potentially eligible participants will be assessed in the ED, or on hospital admission. Assessment of eligibility, recruitment and randomisation should take place as soon as possible (target within 48 hours) after injury. Patients with incapacity who are unable to give informed consent may still be recruited.

Exceptionally, patients who have not been assessed for eligibility at the time of their acute admission, or who were assessed but in whom there was some other delay to study inclusion, may be recruited up to 3 weeks post-injury.

Those who take part will be randomised to continuing in a hard collar for 12 weeks or to early removal of the hard collar.

During the pilot phase, a subset of patients, caregivers and health professionals will be interviewed.

In current standard care, patients with suspected cervical spine injuries are usually (but not universally) immobilised with non-padded trauma collars or blocks, possibly on spinal boards, on admission to the ED. Early removal of this emergency immobilisation and replacement with a padded hard collar (e.g. Miami J, Aspen, Philadelphia) as per standard care is desirable for skin care and comfort. In this study this immobilisation replacement will take place as usual with guidance from ED and spinal service (orthopaedic/ neurosurgical), on-call staff, according to local protocols. This avoids any delay in removal of emergency immobilisation that might be caused by trial procedures to establish eligibility or consent that could lead to poorer quality of care for participants.

All participants will undergo standard care investigations for suspected cervical spine fracture. This includes CT of the cervical spine to identify fractures, and a full neurological examination and assessment. All participants will be discussed with the on-call spinal (neurosurgical/orthopaedic) service unit as per usual protocols. All participants will be given adequate analgesia for neck pain. Participants will only be enrolled following a consultant radiologist report of an odontoid fracture and confirmation from the local spinal consultant that randomisation to non-operative management with or without a hard collar is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Rockwood clinical frailty scale (CFS) of 5 or more, or aged 65 years or over;
* A recent odontoid fracture (type I-III) (within 3 weeks) as assessed on CT, irrespective of degree of fracture angulation, displacement or canal narrowing;
* History of recent trauma (within 3 weeks)
* Determined by spinal consultant (or delegated registrar) as suitable for standard care 12-week treatment with hard collar and for randomisation to treatment without a collar
* Recruited within 3 weeks of injury

Exclusion Criteria:

* New neurological deficit (numbness / weakness) attributable to fracture;
* Assessed as unable to tolerate a hard collar e.g., dystonia, fixed deformity;
* Additional (non-odontoid) cervical spine fracture not suitable for management without a hard collar;
* Underlying condition potentially leading to spinal instability, e.g., ankylosing spondylitis, diffuse idiopathic skeletal hyperostosis (DISH);
* Fracture suspected to be older than three weeks at the time of assessment;
* Consultant spinal surgeon determines fracture requires surgical treatment or is otherwise unsuitable for non-surgical treatment with or without a hard collar;
* If not expected to survive to hospital discharge based on concomitant injuries or illnesses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L Score - (EuroQol five dimensional descriptive system) | 12 weeks
  Primary Outcome is Quality of Life assessed using the EQ-5D-5L questionnaire at 12 weeks post injury. EQ-5D-5L - Is the EuroQol 5D-5L a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

SECONDARY OUTCOMES:
EQ-5D-5L Score - (EuroQol five dimensional descriptive system) | Measured at 2 and 6 weeks and 6 months post injury
  Secondary outcome is Quality of Life assessed using the EQ-5D-5L questionnaire at 2 and 6 weeks and 6 months post injury. EQ-5D-5L - Is the EuroQol 5D-5L a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Neck Disability Index (NDI) | Measured at 2, 6 and 12 weeks and 6 months post injury
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's neck pain related disability. Each question is measured on a scale from 0 (no disability) to 5, and an overall score out of 50 is calculated by adding each item score together. This score is then multiplied by two to give a percentage score. A higher NDI score means the greater a patient's perceived disability due to neck pain.
Numeric Pain Rating Scale (NPRS) | Measured at 2, 6 and 12 weeks and 6 months post injury
  The Numeric Pain Rating Scale is used to measure the patient's perception of their neck pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain imaginable. This data can be collected on paper or over the phone.
Mortality | 6 months post injury
  Mortality
Adverse events | Up to 12 weeks post injury
  Adverse events
Fracture site bony fusion | 12 weeks post injury
  In fracture site bony fusion at approximately 12 weeks assessed on imaging (CT, flexion-extension x-rays or MRI) where performed as part of standard care
Fracture site stability | 12 weeks post injury
  In fracture site stability at approximately 12 weeks assessed on imaging (CT, flexion-extension x-rays or MRI) where performed as part of standard care
Loss of muscle bulk in upper limbs - assessed using a combination of grip strength and muscle bio-impedance | Measured over 12 weeks
  Loss of muscle bulk in upper limbs will be assessed using grip strength and muscle bio-impedance.
  In consenting participants, hand grip strength will be measured using a dynamometer. Participants will be seated, their elbow by their side and flexed to right angles, and a neutral wrist position. The mean of three trials of grip strength will be reported for each hand.
  Bioelectric impedance (Bio-impedance) analysis measurements will be made at the right wrist and ankle, with the subject supine. Muscle mass is calculated according to Janseen et al.
  skeletal muscle mass (kg) =[height2/Bioimepedance x 0.401) +(gender x 3.825) +(age x -0.071)] +5.102
  where height is in centimetres, Bio-impedance in ohms, gender male =1 and female=0, and age is in years. The skeletal muscle index in kg/m2 is obtained by dividing the muscle mass by squared height.
Late injury-related complications | Up to 6 months post injury
  Late injury-related complications, such as new neurological deficit
Total number of hospital admissions or outpatient visits | Up to 6 months post injury
  In patient hospitalisations including outpatient visits and total inpatient bed days
Total amount of health and social care visits/use | Up to 6 months post injury
  Health care, community health and social care use and primary care visits
Compliance with Hard Collar Use | Up to 12 weeks post injury
  Compliance with Hard Collar wear in a sample of patients. iButtons or similar will be placed inside the hard collar of a small sample of patients. These buttons record variations in temperature and can therefore measure compliance with collar wear.
Length of primary admission | The total length of time between a patient's primary admission and their discharge from hospital. Up to 12 weeks after admission.
  Length of primary admission
Discharge destination | Noted at point of discharge of participant. Usually within 12 weeks after admission.
  The location the patient will be discharged to eg. home, care home
Health Economics Analysis | 6 months
  A 6 month within trial analysis will be undertaken based on National Institute for Health and Care Excellence (NICE) reference case recommendations to maximise UK policy relevance. This will include: Adoption of an National Health Service (NHS) and Personal Social Services (PSS) decision perspective; cost-utility approach for primary analysis (results presented in terms of incremental cost per quality adjusted life year (QALY) derived from EQ-5D-5L data with an area under the curve approach, omitting baseline); discount rate of 3.5% for both costs and QALYs (where applicable); and use of probabilistic sensitivity analysis (PSA), to generate cost effectiveness acceptability curves (CEACs). Choice of primary analysis cost per QALY threshold and EQ-5D-5L scoring algorithm will be selected to match NICE preferences. NHS & PSS resource use will be extracted from medical records with some top-up self-report surveying. These will be combined with standard UK price weights to generate costs.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brennan, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient-level data will be available on reasonable request to the Chief Investigator (paul.brennan@ed.ac.uk). The trial protocol and statistical analysis plans will be published and available prior to trial completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The Protocol (and consent form) has been submitted to the British Medical Journal - BMJ Open and will be available once their review is complete.
  The SAP will be available prior to trial completion.
Access Criteria: Available on reasonable request to the Chief Investigator (paul.brennan@ed.ac.uk) as assessed by the study management group

REFERENCES:
- [Derived] Woodfield J, Edlmann E, Black PL, Boyd J, Copley PC, Cranswick G, Eborall H, Keerie C, Khan S, Lawton J, Lowe DJ, Norrie J, Niven A, Reed MJ, Shenkin SD, Statham P, Stoddart A, Tomlinson J, Brennan PM. Duration of External Neck Stabilisation (DENS) following odontoid fracture in older or frail adults: protocol for a randomised controlled trial of collar versus no collar. BMJ Open. 2022 Jul 15;12(7):e057753. doi: 10.1136/bmjopen-2021-057753. PMID 35840308